CLINICAL TRIAL: NCT02477488
Title: Optimal Administration of Allopurinol in Dialysis Patients : A Chronotherapy Trial
Brief Title: Optimal Administration of Allopurinol in Dialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Michel Vallée, Nephrologist, M.D., Ph.D., FRCP(C), Maisonneuve-Rosemont Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 14106
Record Dates: First submitted 2015-06-17; First posted 2015-06-22 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Gout; Renal Insufficiency
Keywords: Allopurinol; Renal Dialysis
MeSH Terms: conditions — Gout; Renal Insufficiency | interventions — Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Allopurinol HS (Experimental): Allopurinol at bedtime compared to AM administration
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Drug: Allopurinol — Administration of allopurinol is changed to bedtime (hs) for each patient, at the same dosage as was previously prescribed.
  Other Names: Zyloprim

SUMMARY:
Gout has a strong association with the metabolic syndrome, and it is often seen in patients with renal insufficiency. Allopurinol is a medication intended to lower uric acid and therefore prevents gout attacks. Its metabolism is mainly renal, and some evidence shows that it is also dialyzable. The hypothesis is that allopurinol would be more efficacious to lower uric acid if it was given after dialysis only. The investigators will then switch administration of allopurinol to bedtime for dialysis patients currently taking that medication.

DETAILED DESCRIPTION:
Gout has a strong association with the metabolic syndrome, and it is often seen in patients with renal insufficiency. A study has shown an incidence of fifteen percent of gout in the first five years spent in dialysis and it was associated with an increased mortality. Allopurinol is a medication intended to lower uric acid and therefore prevents gout attacks. Its metabolism is mainly renal, and some studies from the early 1960s demonstrated that it is also dialyzable. At the moment, we do not have strong evidence of the optimal dosage of allopurinol with modern techniques of dialysis. The hypothesis is that allopurinol would be more efficacious to lower uric acid if it was given after dialysis only. The investigators will then switch administration of allopurinol to bedtime for dialysis patients currently taking that medication. Dosage of uric acid will be performed to assess the efficacy of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who receive chronic treatments of hemodialysis at Maisonneuve-Rosemont Hospital
* Subjects who take allopurinol for at least a month

Exclusion Criteria:

* Subjects who have had an acute gout attack in the past month
* Subjects with tumor lysis syndrome
* Sujects who have a history of hypersensitivity reaction to allopurinol
* Subjects with hepatic insufficiency
* Women who are pregnant or planning to become pregnant in the next three months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in uric acid levels from baseline | 6 weeks
  Compare the efficacy of allopurinol when given before versus after dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Michel Vallée, MD, PhD, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Cohen SD, Kimmel PL, Neff R, Agodoa L, Abbott KC. Association of incident gout and mortality in dialysis patients. J Am Soc Nephrol. 2008 Nov;19(11):2204-10. doi: 10.1681/ASN.2007111256. Epub 2008 May 28. PMID 18508965